CLINICAL TRIAL: NCT00695942
Title: Prediction of the Risk of Placental Vascular Pathology and Venous Thromboembolic Disease: Role of Angiogenic Factors, Hemostasis and Uterine Artery Doppler
Brief Title: Prediction of the Risk of Placental Vascular Pathology and Venous Thromboembolic Disease
Acronym: AngioPred
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: ARGOS (Unknown); Association de la Vallée de l'Ondaine (Unknown)
Responsible Party: Sponsor
Other Study IDs: 0708115; 2007-A01448-45; DGS 2008-0167
Record Dates: First submitted 2008-06-05; First posted 2008-06-12 (Estimated); Last update posted 2012-05-17 (Estimated); Status verified 2012-05

CONDITIONS: Placental Vascular Pathologies; Venous Thromboembolism Diseases
Keywords: preeclampsia; eclampsia; retroplacental hematoma; vascular IUGR; IUFD; VTE
MeSH Terms: conditions — Pre-Eclampsia; Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma and serum samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: pregnancy women

SUMMARY:
Venous thromboembolic (VTE) disease is the first cause of maternal mortality in the world. Some other pregnancy pathologies called Placental Vascular Pathologies (PVP) are linked to VTE by biological thrombophilia and are the principal cause of perinatal mortality. the identification of predictive factors of risk of occurrence or recurrence of two pathologies could enable us to propose an appropriate monitoring of patients at risk.

DETAILED DESCRIPTION:
Main aim: To evaluate echographic, doppler and biological markers in a prospective manner as a potential predictive factor of risk of PVP and VTE.

ELIGIBILITY:
Inclusion Criteria:

* previous history of one or more PVC episodes (preeclampsia, HELLPs, retroplacental hematoma, vascular IUGR<10th percentile, recurrence miscarriage >2, unexplained IUFD or IUFD after abruption placentae, eclampsia.
* Previous history of personal VTE
* Diabete (treated with diet or insulin)
* chronic hypertension
* chronic renal pathology
* lupus
* obesity
* Antihopholipids syndrome
* early and late pregnancy (<18 years, >38 years)
* family history of cardiovascular disease of VTE
* known biological thrombophilia without any personal past history of PVC or VTE

Exclusion Criteria:

* Multiple pregnancy
* past history of in utero fetal death due to congenital malformations, rhesus incompatibility or an infection
* previous history of IUGR which etiology was a chromosomal, genic or infectious anomaly

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2008-06; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
sFlt1/plGF ratio | 20, 24, 28, 32, 36 weeks

SECONDARY OUTCOMES:
SFlt1/PlGF ratio as predictive threshold to develop a PVP and/or a VTE | 20, 24, 28, 32, 36 SA
thrombin generation test (TGT) as potential predictive factor risck oj PVP and VTE | 20, 24, 28, 32 and 36 weeks
sEng, rTFPI, D-Dimer, uCRP, PP13 as potential predictive factor of risk of PVP and or VTE | 20, 24, 28, 32 and 36 weeks
echographic data as potential predictive factors of VTE and or PVP | 22 and 32 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Céline CHAULEUR, MD, Principal Investigator — CHU de Saint-Etienne
Locations (3):
- France (3):
  - Service d'Hématologie - CHU de Nîmes, Nîmes
  - Service de gynécologie Obstétrique, Nîmes
  - Service de Gynécologie Obstétrique - CHU Saint-Etienne, Saint-Etienne